CLINICAL TRIAL: NCT04186221
Title: Continued Access Protocol To Evaluate the Effectiveness of the Portable Organ Care System (OCS) Liver for Preserving and Assessing Donor Livers for Transplantation.
Brief Title: OCS Liver PROTECT Continued Access Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LVR10202019
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplant

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, continued access protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: OCS Liver System

INTERVENTIONS:
Device: OCS Liver System — OCS Liver System for preserving and assessing donor livers for transplantation

SUMMARY:
Continued Access Protocol to evaluate the effectiveness of the OCS Liver System to preserve and assess donor livers.

DETAILED DESCRIPTION:
A prospective, single arm, continued access protocol to evaluate the effectiveness of the OCS Liver System to preserve and assess donor livers having one or more of the following characteristics:

1. Donor age equal to or greater than 40 years old, or
2. Expected cross clamp time of 6 hours or greater, or
3. Donor after circulatory death (DCD) with age less than or equal to 55 years; or
4. Steatotic lever >0% and less than or equal to 40% at time of retrieval, based on pre-retrieval histology)

A maximum of 21 sites will enroll up to 184 transplanted liver recipients. The primary effectiveness endpoint will be the incidence of Early Allograft Dysfunction (EAD) or primary non-function.

All recipients will be followed for 24 months from the date of transplantation (some of which will be post-market).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Registered primary liver transplant candidate, male or female
* Age ≥ 18 years
* Signed (1) written informed consent document and (2) authorization to use and disclose protected health information

Exclusion Criteria:

* Acute, fulminant liver failure
* Prior solid organ or bone marrow transplant
* Chronic use of hemodialysis or diagnosis of chronic renal failure, defined as chronic serum creatinine of > 3 mg/dl for > 2 weeks and/or requiring hemodialysis
* Multi-organ transplant
* Ventilator dependent
* Dependent on > 1 IV inotrope to maintain hemodynamics

Donor Inclusion Criteria

* Donor age ≥ 40 years, or
* Expected cross-clamp time ≥ 6 hours, or
* Donor after circulatory death (DCD) with age ≤ 55 years, or
* Steatotic liver > 0% and ≤ 40% macrosteatosis at time of retrieval

Donor Exclusion Criteria

* Living donors
* Liver intended for split transplants
* Positive serology (HIV, Hepatitis B surface antigen & Hepatitis C)
* Presence of moderate or severe traumatic liver injury, or anatomical liver abnormalities that would compromise ex-vivo perfusion of the donor liver (i.e., accessory blood vessels or other anatomy that require surgical repair) and livers with active bleeding (e.g., hematomas)
* Donor livers with macrosteatosis of > 40% based on retrieval biopsy readout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elbetanony, MD, Study Director — TransMedics
Locations (17):
- United States (17):
  - Scripps, La Jolla, California
  - University of California San Diego, La Jolla, California
  - UCSF, San Francisco, California
  - Tampa General, Tampa, Florida
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Montefiore Einstein Center for Transplantation, The Bronx, New York
  - Ohio State University, Columbus, Ohio
  - Methodist University Hospital, Memphis, Tennessee
  - University of Texas Southwest, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia

REFERENCES:
- [Derived] Kubal C, Mihaylov P, Holden J. Oncologic indications of liver transplantation and deceased donor liver allocation in the United States. Curr Opin Organ Transplant. 2021 Apr 1;26(2):168-175. doi: 10.1097/MOT.0000000000000866. PMID 33650998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 74
Completed (Completing the 30 day visit.) | 73
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.01 (11.572)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 62
  More than one race | 0
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Participants With Early Liver Allograft Dysfunction (EAD)
Description: Participants with Early liver Allograft Dysfunction (EAD) or primary non-function, defined as presence of one or more of the following criteria: AST level > 2000 IU/ml within the first 7 postoperative days; Bilirubin ≥ 10 mg/dl on postoperative day 7; INR ≥ 1.6 on postoperative day 7; or Primary non-functioning graft within the first 7 days (defined as irreversible graft dysfunction requiring emergency liver re-transplantation or death, in the absence of immunologic or surgical causes)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 74
Participants | 19

2. Secondary Outcome: Patient Survival at Day 30 After Transplant
Description: Patient survival at day 30 post transplantation.
Time Frame: 30 days after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 74
Participants | 73

ADVERSE EVENTS:
Time Frame: Liver graft-related serious adverse events (LGRSAEs) were collected up to the 30-day follow-up after transplantation for the safety endpoint. All-cause mortality is reported through 30-days post transplant.
Description: Only death and serious adverse events were assessed.
  Other (Not Including Serious) Adverse Events were not monitored/assessed, and therefore are not reported.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 1/74
Serious Adverse Events (participants affected / at risk) | 4/74
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=74)
Hepatic artery thrombosis (Hepatobiliary disorders) | 3 (3)
Hepatic artery stenosis (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sites shall have right to publish results. To balance this right with TransMedics' (TM) proprietary interests, site will submit manuscripts intended for publication for TM review at least 30 days prior to submission date. TM will complete its review within 30 days of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT04186221/Prot_SAP_000.pdf